CLINICAL TRIAL: NCT03653052
Title: CALIBRATION: An Exploratory Study in Patients With Advanced Oesophageal Malignancies Receiving MEDI4736 (Durvalumab), Investigating Whether Early Changes in Circulating Tumour DNA Can Predict Tumour Response
Brief Title: Do Changes in ctDNA Predict Response for Patients With Oesophageal Cancer Receiving Durvalumab
Acronym: CALIBRATION
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Simon C Pacey, MD (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Simon C Pacey, MD, Chief Investigator, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALIBRATION
Record Dates: First submitted 2018-07-09; First posted 2018-08-31 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Oesophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Durvalumab (Experimental): Patients with advanced oesophageal cancer will be administered with 1500mg of durvalumab once every 4 weeks for up to 6 months.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab will be administered via an infusion in the arm, over a duration of up to 1 hour.
  Other Names: MEDI4736

SUMMARY:
Patients with cancer are increasingly being treated with drugs designed to modulate the response of their immune system, broadly to boost their body's defences against cancer. However, there is an unmet need to identify which patients are unlikely to benefit. Deciding on benefit from therapy uses standard imaging methods (e.g. CT scans), which can take time (months) whereas DNA in the bloodstream could be measured more rapidly.

The main aim of this study is to assess whether changes in the level of circulating tumour DNA (ctDNA) can quickly determine a patients response. This would enable patients to change therapies more quickly if they are not responding and reduce exposure to unnecessary side effects.

DETAILED DESCRIPTION:
Measuring circulating (plasma) tumour DNA has been described as a 'liquid biopsy' able to study a tumour without invasive biopsy. By measuring ctDNA at different time points the investigators can detect tumour changes that indicate if the patient is responding to treatment or not.

This trial has been designed as a prospective, open label, non-randomised trial where patient with advanced oesophageal cancer will be treated with MEDI4736 (durvalumab), a drug designed to alter the immune system response. Samples will be taken to regularly to measure ctDNA levels and compared to patients response at 6 months when undergoing standard CT scans.

The study will run at a single centre (Addenbrookes Hospital, Cambridge). Nineteen, evaluable, patients will receive durvalumab until progression while detailed studies will assess their tumour and immune response.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent to participate
* Aged ≥ 18 years at time of consent
* Confirmed advanced oesophageal cancer for which the patient must have received at least one prior line of standard of care treatment
* Predicted life expectancy ≥ 3 months
* Eastern Cooperative Oncology Group (ECOG) PS 0 or 1
* Measurable disease, as defined by RECIST v1.1.
* In the investigator's opinion, have an accessible and biopsiable tumour lesion for additional research biopsy, to which the patient will have to consent at screening.
* Adequate hematologic and organ function, defined by:

  * ANC ≥ 1500 cells/μL (no GCSF support 2 weeks prior to trial entry)
  * Platelet count ≥ 100,000/μL
  * Haemoglobin ≥ 9.0 g/dL
  * AST or ALT ≤ 2.5 times the upper limit of normal (ULN), (except patients with documented liver metastases where AST and/or ALT can be ≤ 5×ULN)
  * Serum bilirubin ≤1.5 × ULN. (Except patients with confirmed Gilbert's syndrome)
  * INR and APTT ≤ 1.5×ULN.
  * Calculated creatinine clearance (CrCl) ≥ 40 mL/min (Cockcroft-Gault formula)
* Negative pregnancy test in women of child-bearing potential or evidence of postmenopausal status

Exclusion Criteria:

* Weight of ≤30kg
* Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment.
* Participation in other clinical trials involving active treatment for the malignant disease.
* Received radiotherapy treatment on a wide body field, or an equivalent to more than 30% of the bone marrow, within the last 4 weeks.
* Any unresolved symptom NCI CTCAE Grade ≥2 from previous anticancer therapy (with the exception of alopecia and vitiligo).
* Active or prior documented autoimmune or inflammatory disease (except vitiligo) within the last 3 years, for example:

  * Intestinal: Inflammatory Bowel Disease (Colitis, Crohn's Disease), Diverticulitis (with the exception of Diverticulosis), Coeliac Disease, Irritable Bowel Disease
  * Vascular: any type of Vasculitic disorder, i.e.: Wegner syndrome.
  * Endocrine: any endocrine alteration related to an auto-immune process i.e.: Hashimoto syndrome. NOTE: patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement treatment may be included at the discretion of the CI.
  * Respiratory: Active Pneumonitis (of any origin: inflammatory or infectious), Sarcoidosis.
  * Dermatological: Psoriasis, Lupus/SLE.
  * Other: Rheumatoid Arthritis, Hypophysitis, Uveitis.
* History of organ transplant that requires use of immunosuppressive medications or any medical condition in which immunosuppressive agents were administered, including but, not limited to:

  * Systemic corticosteroids.
  * Methotrexate, azathioprine
  * Tumour necrosis factor alpha (TNF-α) blockers
* History of active primary immunodeficiency.
* Receipt of live, attenuated vaccine within the last 30 days.
* Other invasive malignancy within the last 3 years. Patients with previous history of malignancies with a negligible risk of metastasis or death and treated with expected curative intent are eligible at the investigator's discretion, for example:

  * Carcinoma in situ of the cervix
  * Basal or squamous cell skin cancer
  * Localized low to intermediate risk prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse; or prostate cancer (Stage T1/T2a, Gleason ≤ 6 and PSA < 10 ng/mL) undergoing active surveillance and treatment naive
* Women who are pregnant or lactating/ breast feeding.
* Male or female patients with reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab.
* Uncontrolled intercurrent illness, including but not limited to, on-going or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Brain metastases unless asymptomatic, treated and stable and not requiring steroids in the last 4 weeks. Patients with known or suspected brain metastases at screening should have a CT/ MRI of the brain prior to trial entry.
* History of leptomeningeal carcinomatosis.
* Active infection or use of antibiotics (ATB) 14 days prior to Cycle 1 Day 1 of treatment. Patients receiving prophylactic treatment are eligible.
* Active infection including tuberculosis (clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or known human immunodeficiency virus (positive HIV1/2 antibodies).

  * Subjects with a past or resolved HBV infection (defined as: presence of hepatitis B core antibody -anti-HBc- and absence of hepatitis B surface antigen -HbsAg-) are eligible.
  * Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Major surgical procedure (investigator defined) within 4 weeks prior to first dose or anticipation of the need for a major surgical procedure during the course of the trial other than for diagnosis.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to durvalumab or any of its excipients, chimeric or humanized antibodies or fusion proteins.
* Patients previously treated with immune (checkpoint inhibition) therapy
* Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical trial due to safety concerns, compliance with clinical trial procedures or interpretation of trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Clinical response to therapy (durvalumab) | 26 weeks
  Changes in ctDNA levels (from baseline to C1/C2) compared with objective RECIST radiological response at 26 weeks

OTHER OUTCOMES:
Immunological milieu in tumour samples | 33 months
  Changes in intra-tumoural T-Cell distribution, immunostaining and other biomarkers of immune activation following exposure to durvalumab
ctDNA/plasma sampling | 33 months
  Tracking immunological changes and variability in immune-cells (clonality, T-cell receptor, tumour infiltrating lymphocytes) and neoantigens; tumour specific mutation(s); and, blood-based biomarkers following exposure to durvalumab
ctDNA's potential to identify tumour resistance mechanisms | 33 months
  Tracking immunological changes and variability in immune-cells (clonality, T-cell receptor, tumour infiltrating lymphocytes) and neoantigens; tumour specific mutation(s); and, blood-based biomarkers following exposure to durvalumab
Correlation in ctDNA levels and occurrence of clinically related adverse events | 33 months
  Variations in tumour variant alelle frequencies (VAF) compared with the occurrences of >= Grade 2 treatment related side effects
Integrate the use of iRECIST criteria | 33 months
  Compare responses by RECIST and iRECIST criteria
Patient stratification according to predefined genetic signatures | 33 months
  Time taken and costs incurred from sample collection through to the generation of data and, the correlation between response to durvalumab and the genetic signature that the patient is assigned to
Ex-vivo effect of compounds on tumour/cell models | 33 months
  Ex-vivo response to durvalumab using patient derived model systems

CONTACTS AND LOCATIONS:
Overall Officials: Simon Pacey, Principal Investigator — Cambridge University Hospitals
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom